CLINICAL TRIAL: NCT06652360
Title: A Pilot Study to Investigate the Relative Effectiveness and Safety of Chemical Wound Debridement and Curettage in the Treatment of Venous and Mixed Aetiology Leg Ulcers.
Brief Title: Chemical Debridement and Leg Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DEBx Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCHEM2023_VLU
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Venous Leg Ulcers; Mixed Ulcer
Keywords: chemical debridement; mechanical debridement; topical dessicating agent; venous leg ulcer; chronic wound
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemical Debridement (Active Comparator): 1 single treatment of chemical debridement will be applied in this arm at initiation visit. No repeated treatment done in this trial
  Interventions: Device: Chemical Debridement
- Sharp debridement (Active Comparator): In the control arm wound debridement by curettage will be performed at initiation visit and after 2 weeks when clinician deems this necessary, conform standard of care protocol
  Interventions: Device: Curettage debridement

INTERVENTIONS:
Device: Chemical Debridement — The chemical debridement is a dehydrating agent in a gel shape that will dry out the woundbed and biofilm.
  Arms: Chemical Debridement
Device: Curettage debridement — The use of a currette will clean the wound bed. Debridement by mechanically removing the necrotic tissue and biofilm. This is performed confrom the standard of care standards.
  Arms: Sharp debridement

SUMMARY:
A pilot study to investigate the relative effectiveness and safety of chemical wound debridement and curettage in the treatment of venous and mixed aetiology leg ulcers.

DETAILED DESCRIPTION:
A pilot study to investigate the relative effectiveness and safety of chemical wound debridement versus the curettage wound debridement in the treatment of venous and mixed aetiology leg ulcers in the United Kingdom

ELIGIBILITY:
Inclusion Criteria:

* Participants with a venous leg ulcer or mixed aetiology ulcer.
* Duration of wound ≥ 6 weeks ≤ 5 years
* Wound is ≥ 5 cm2 ≤ 200cm2
* Presence of at least 25% visible slough within the wound bed
* The Participant must be able to understand the study and provide written informed consent
* No clinical signs of infection

Exclusion Criteria:

* Known hypersensitivity or contraindications to any of the wound treatments, dressings or compression bandaging to be used in the trial
* Current local or systemic antibiotics in the week prior to inclusion
* Clinically infected wound as determined by the presence of 3 or more of the following clinical signs: perilesional erythema, pain between two dressing changes, malodorous wound, abundant exudate and oedema
* Prolonged treatment with immunosuppressive agents or high dose corticosteroids
* Participants who have a current illness or condition which may interfere with wound healing in the last 30 days (carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse)
* Participants who have participated in a clinical trial on wound healing within the past month
* Participants with a known history of non- adherence with medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Wound surface | 12 weeks
  Change in wound surface area (cm^2)
Wound Debris | 12 weeks
  Change in the percentage of the wound bed covered with slough

SECONDARY OUTCOMES:
Wound healing | 12 weeks
  Number of healed wounds, according BWAT score ranging from 13 (minimal) - 65 (extreme severity)
wound condition | 12 weeks
  Condition of the wound bed by percentage of granulation tissue, percentage covered in slough, exudate; Measured via visual assessment totalling up to 100% (e.g. 30% granulation, 25% slough, 25% necrosis, 20% exudate)
Quality of Life | 12 weeks
  Health-related quality of life assessed using WoundQOL (an established validated questionair production a single number between 0-1 with 1 being the optimal quality of life)
Patient Comfort in treatment process | 12 weeks
  Pain measured Participant pain measured using Visual Analogue Scale (VAS 0-10, 0 being painless and 10 being most pain to be imagined)
Device Safety | 12 weeks
  Incidence of Treatment-related Adverse Events Incidence of Adverse Events of Special Interest
Treatment Comfort in performance and acceptance | 12 weeks
  Participant and staff acceptance of the debridement methods by questionnaire. Score denoted in precentage with 100% being fully comfortable and accepted.
wound condition | 12 weeks
  Condition of peri-ulcer skin and surrounding skin (healthy, bumpy, integrated, fragile))
wound condition | 12 weeks
  Maloudour (yes, no);

CONTACTS AND LOCATIONS:
Locations (1):
- Pioneer wound healing and lymphedema centres, Eastbourne, United Kingdom